CLINICAL TRIAL: NCT06822959
Title: Pharmacogenetics, Therapeutic Drug Monitoring (TDM) and Active Pharmacovigilance as Innovative Tools Aimed at the Optimisation/ Appropriateness of Drug Therapy and the Minimisation of the Risks of ADRs in Clinical Practice: a Multidisciplinary Approach Exportable at National Level
Brief Title: Pharmacogenetics, Therapeutic Drug Monitoring (TDM) and Active Pharmacovigilance as Innovative Tools Aimed at the Optimisation/ Appropriateness of Drug Therapy
Status: Recruiting | Type: Observational
Sponsor: Direzione centrale salute, politiche sociali e disabilità (Other)
Collaborators: Centro di Riferimento Oncologico - Aviano (Other); IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2022-14
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Adverse Drug Reaction (ADR)
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adult patients: Adult cancer patients
  Interventions: Other: Pharmacogenetics, TDM and MedReview
- Pediatric patients: Pediatric patients with chronic inflammatory diseases
  Interventions: Other: Pharmacogenetics, TDM and MedReview

INTERVENTIONS:
Other: Pharmacogenetics, TDM and MedReview — Patients will undergo pharmacogenetics, TDM and MedReview analyses according to the study protocol

SUMMARY:
The primary goal of this observational study is to evaluate the feasibility of implementing a multidisciplinary approach based on pharmacogenetics, TDM (Therapeutic Drug Monitoring) and MedReview into the clinical practice in order to optimize the appropriateness of drugs prescription and to minimise the risk of Adverse Drug Reactions (ADRs) in adult cancer patients and in pediatric patients affected by chronic inflammatory diseases. This approach of active pharmacovigilance will also allow a better definition of the causality assessment of ADRs through the direct implementation of data quality in the reporting forms. The study may therefore constitute an example of an approach for both the prevention of ADRs and the optimization of drug use, and for the integration of pharmacogenetics, TDM, and the MedReview data into the National Pharmacovigilance Reports for an improved and innovative evaluation of adverse events, aiming at the implementation of this approach in the regional context.

DETAILED DESCRIPTION:
Primary aim of the study:

To implement the use of pharmacogenetics, TDM, and MedReview at the regional level supporting their utility through an observational approach to assess the effects of these innovative methods, already active in IRCCS, for the optimization of appropriate drug use and minimization of ADR risk in adult and pediatric oncology patients, as well as pediatric patients with chronic inflammatory diseases. Specifically, the aim is to evaluate the incidence of ADRs in patients treated based on pharmacogenetics, TDM, and MedReview compared to historical cases treated according to the standard of care before the implementation of the proposed innovative methodologies.

Secondary aims of the study:

1. To evaluate the "Causality Assessment" between ADR and drug based on the enhanced data quality deriving from the integration of pharmacogenetics, TDM and MedReview into the Pharmacovigilance report.
2. To propose the systematic integration of the results related to pharmacogenetics, TDM, and MedReview within the existing fields of the current ADR reporting form. This aims to develop a proposal for updating AIFA procedures related to the inclusion of this type of evidence-based information in the National Pharmacovigilance Network (RNF), with a potential update of the reporting form.

ELIGIBILITY:
Inclusion Criteria:

Patients who are candidates for therapy with:

* Abemaciclib,
* Palbociclib,
* Ribociclib,
* Letrozole,
* Tamoxifen,
* Olaparib,
* Niraparib,
* Rucaparib,
* Imatinib,
* Sunitinib,
* Sorafenib,
* Regorafenib,
* Lenvatinib,
* Irinotecan,
* Capecitabine,
* 5-Fluorouracil,
* Infliximab,
* Cyclophosphamide,
* Methotrexate,
* Adalimumab,
* 6-Mercaptopurine/Azathioprine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are candidates for therapy with: Abemaciclib, Palbociclib, Ribociclib, Letrozole, Tamoxifen, Olaparib, Infliximab, Cyclophosphamide, Methotrexate, Irinotecan, Capecitabine, 5-Fluorouracil, Noraparib, Adalimumab, Imatinib, Regorafenib, Lenvatinib, Sorafenib, Sunitinib, Rucaparib, 6-MP/ Azathioprine
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Patients treated with study drugs tested with pharmacogenetic and TDM analysis | Up to 2 years
  Percentage of patients treated with study drugs tested with pharmacogenetic and TDM analysis on total patients treated
MedReview reports | Up to 2 years
  Number of MedReview reports
ADRs in patients treated on the basis of pharmacogenetics, TDM and MedReview | Up to 2 years
  Incidence of ADRs in the study cohorts
Comparison of ADRs in patients treated on the basis of pharmacogenetics, TDM and MedReview and retrospective data | Up to 2 years
  Difference in incidence of ADRs in the prospective cohort will be tested against historical data with binomial test

SECONDARY OUTCOMES:
Integration of pharmacogenetics, TDM and MedReview information in the existing tool for the evaluation of "Causality assessment" between ADR and specific drug | Up to 2 years
  Change of Causality Assessment. The change is evaluated as the number of "definite" and "probable" associations between ADRs and suspected drugs compared with historical data
Proposal for updating the pharmacovigilance reporting forms including Pharmacogenetics, TDM and MedReview information in the National Network of Pharmacovigilance | Up to 2 years
  Frequencies of new reports sent to the National Pharmacovigilance Network, including pharmacogenetics, TDM, and drug interaction data
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 v3 | Up to 2 years
  The EORTC QLG Core Questionnaire (EORTC QLQ-C30) is a 30-item instrument designed to measure quality of life in all cancer patients.
  The possible answers to the questionnaire range from a minimum value ("not at all") to a maximum value ("very much"). Higher values indicate a worse quality of life.
  Mean and standard deviation of scores at EORTC QLQ-C30 v3 questionnaire will be evaluated.
Costs of ADRs management | Up to 2 years
  Median and interquartile range of costs
Concordance between plasmatic concentration measured with conventional methods and with new methods such as Dried Blood Spot (DBS) | Up to 2 years
  Lin's correlation coefficient between plasmatic concentration and DBS estimation
Correlation between pharmacogenetic profile and drug exposure (TDM) | Up to 2 years
  Difference in drug exposure measured as Cmin for different pharmacogenetic profiles
Correlation between ADRs, TDM and pharmacogenetics analyses | Up to 2 years
  Frequencies of ADRs in different subgroups of patients defined by TDM and pharmacogenetic profiles
Correlation between ADRs, TDM and pharmacogenetics analyses | Up to 2 years
  Frequencies of severe ADRs in different subgroups of patients defined by TDM and pharmacogenetic profiles

CONTACTS AND LOCATIONS:
Overall Officials: Erika Cecchin, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (2):
- Italy (2):
  - Centro di Riferimento Oncologico di Aviano (CRO), Aviano, Pordenone
  - IRCCS materno infantile Burlo Garofolo di Trieste, Trieste, Trieste

IPD SHARING:
Plan to Share IPD: No